CLINICAL TRIAL: NCT04531085
Title: Multi-center Comparative Study of Operative Vs Nonoperative Treatment of Medial Epicondyle Fractures in Children and Adolescents
Brief Title: Treatment of Medial Epicondyle Fractures in Children and Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Petra Grahn, Hand Surgeon, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HUS/1443/2019
Record Dates: First submitted 2020-08-22; First posted 2020-08-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Medial Epicondyle Fracture of the Humerus; 7 To16 Year Old Children and Adolecents; More Than 2 Mm of Displacement

STUDY DESIGN:
Intervention Model Description: Non-inferiority RCT 1:1 ratio
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- RCT operative (Active Comparator): Procedure of preference is open reduction and internal fixation (ORIF) with cannulated non-resolvable 4.0mm screw with or without washer. If the fracture fragment is too small or fragmented for screw fixation 1.6mm - 1.8mm Kirshner-wires and/or bone anchor are used. Long arm cast for 4 weeks.
  Interventions: Procedure: Operative treatment
- RCT Non-operative (Active Comparator): Non-operative treatment means upper limb immobilization with forearm in neutral pro-supination with a long arm cast for 4 weeks.
  Interventions: Procedure: Long arm cast
- Patient preference operative (Other): Procedure of preference is open reduction and internal fixation (ORIF) with cannulated non-resolvable 4.0mm screw with or without washer. If the fracture fragment is too small or fragmented for screw fixation 1.6mm - 1.8mm Kirshner-wires and/or bone anchor are used. Long arm cast for 4 weeks.
  Interventions: Procedure: Operative treatment
- Patient preference non-operative (Other): Non-operative treatment means upper limb immobilization with forearm in neutral pro-supination with a long arm cast for 4 weeks.
  Interventions: Procedure: Long arm cast

INTERVENTIONS:
Procedure: Operative treatment — Surgery
  Arms: Patient preference operative; RCT operative
Procedure: Long arm cast — cast immobilization
  Arms: Patient preference non-operative; RCT Non-operative

SUMMARY:
Cast immobilization in situ versus open reduction and internal fixation of displaced medial epicondyle fractures in children between 7 and 16 years old. A non-inferiority randomized controlled trial.

DETAILED DESCRIPTION:
This is a multicenter, controlled, prospective, randomized non-inferiority study comparing operative treatment to non-operative treatment of over 3 mm dislocated pediatric medial epicondyle fractures without joint incarceration or ulnar nerve dysfunction. A total of 120 patients will be randomized in 1:1 ratio to either operative or non-operative treatment. The study will have a parallel non-randomized patient preference arm. Non-operative treatment will be upper limb immobilization with long arm cast for 4 weeks. Operative treatment will be open reduction and internal fixation (ORIF). Data is collected at baseline and at each follow-up up to 2 years. Quick-DASH is used as primary outcome measure. Secondary outcomes are patient reported pain, differences in range of motion, PedsQL Life inventory questionnaire as well as Mayo elbow preformance score.

ELIGIBILITY:
Inclusion Criteria:

- Over 2 mm displaced medial epicondyle fracture of humerus on primary AP or lateral X-ray

Exclusion Criteria:

* Ulnar nerve dysfunction
* Pathological fracture
* Open fracture
* Systemic bone disease
* Concomitant fracture or injury of the same upper limb requiring operative intervention
* Other disease preventing participation in full follow-up regime or range of motion exercises

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2019-08-30 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Quick Disabilities of the Arm, Shoulder and Hand score questionnaire(QuickDASH) | 12 months
  Minimum value is 0 and maximum 100. Higher value indicates worse function. Statistically significant difference in QuickDASH score is 6.8 (18) at 12 months FU.

SECONDARY OUTCOMES:
Range of Motion (ROM) degrees difference of the elbow as compared to uninjured arm | 12 months
  Difference in active ROM in comparison to uninjured arm. Maximum value is 160 degrees minimum 0. Lower value indicates better outcome.
Measurement Model for the Pediatric Quality of Life Inventory questionnaire (PedsQL) | 12 months
  Minimum score is 0 and maximum 100. Higher score indicates better health related quality of life.
Measurement Model for the Pediatric Quality of Life Inventory Pediatric Pain Questionaire (PEDS QL PPQ) | 12 months
  Minimum score 0 maximum 10. Higher value indicates higher pain intensity.
Cosmetic Visual Analoque Scale (CVAS) | 12 months
  Minimum score 0 maximum 100. Higher value indicates better cosmetic appearance
Mayo Elbow Performance Score (MEPS) | 12 months
  Minimum score 0 maximum 100. Higher value indicates better performance.
Need for additional procedures (number) | 12 months
  Minimum value 0, no maximum value. Lower value indicates better outcome.
Grip strength (kg) with hand held dynamometer (jamar) | 12 months
  compared to standard for age kg/age
Sensation and cold intolerance | 12 months
  semmes-weinstein monofilaments scored as normal or abnormal

CONTACTS AND LOCATIONS:
Overall Officials: Petra Grahn, MD, Principal Investigator — Helsinki University Hospital, New Childrens Hospital
Locations (4):
- Finland (4):
  - HUS New Childrens Hospital, Helsinki
  - Kuopio University Hospital, Kuopio
  - Oulu University Hospital, Oulu
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request. Any requests should be sent to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: upon request. Most of the above published in BMJ Open.
Access Criteria: Please see BMJ open
URL: https://bmjopen.bmj.com/content/11/5/e044627

REFERENCES:
- [Derived] Grahn P, Helenius I, Hamalainen T, Kivisaari R, Nietosvaara Y, Sinikumpu JJ, Jalkanen J, Loyttyniemi E, Ahonen M; Finnish Pediatric Orthopedic Study Group Investigators. Casting vs Surgical Treatment of Children With Medial Epicondyle Fractures: A Randomized Clinical Trial. JAMA Netw Open. 2025 May 1;8(5):e258479. doi: 10.1001/jamanetworkopen.2025.8479. PMID 40327343
- [Derived] Hamalainen T, Ahonen M, Helenius I, Jalkanen J, Lastikka M, Nietosvaara Y, Salonen A, Sinikumpu JJ, Grahn P. Cast immobilisation in situ versus open reduction and internal fixation of displaced medial epicondyle fractures in children between 7 and 16 years old. A study protocol for a randomised controlled trial. BMJ Open. 2021 May 3;11(5):e044627. doi: 10.1136/bmjopen-2020-044627. PMID 33941629
- See also: Protocol publication — https://bmjopen.bmj.com/content/11/5/e044627